CLINICAL TRIAL: NCT04735770
Title: Laparoscopically Inserted Transversus Abdominis Plane Block Versus Wound Local Anesthesia in Laparoscopic Endometriosis Surgery: a Prospective Randomized Controlled Double-blinded LTAP-trial
Brief Title: LTAP Block in Endometriosis Surgery - a Randomised Controlled Double-blind Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Anna Terho, Principal Investigator, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OuluUH/Urogyn
Record Dates: First submitted 2021-01-19; First posted 2021-02-03 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Endometriosis; Peritoneum; Postoperative Pain
Keywords: endometriosis; postoperative pain management; laparoscopic surgery; gynecological surgery
MeSH Terms: conditions — Endometriosis; Pain, Postoperative | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTAP (Experimental): Patients receive laparoscopically inserted TAP block with levobupivacain and local wound anesthesia injections with saline.
  Interventions: Procedure: Postoperative pain management: LTAP block or local wound anesthesia with levobupivacaine
- Local wound analgesia (Active Comparator): Patients receive laparoscopically inserted TAP block with saline and local wound anesthesia injections with levobupivacaine.
  Interventions: Procedure: Postoperative pain management: LTAP block or local wound anesthesia with levobupivacaine

INTERVENTIONS:
Procedure: Postoperative pain management: LTAP block or local wound anesthesia with levobupivacaine — Postoperative pain management

SUMMARY:
The purpose of this study is to compare the efficacy and safety of laparoscopically inserted transversus abdominis plane block (LTAP) in comparison to local wound analgesia in laparoscopic surgery due to suspected or diagnosed peritoneal endometriosis.

DETAILED DESCRIPTION:
The LTAP-trial is a prospective randomized controlled double-blinded study comparing the efficacy and safety of LTAP with local wound analgesia in laparoscopic endometriosis surgery. Patients are randomized to receive LTAP with levobupivacain and wound infiltration with placebo or wound infiltration with levobupivacain and LTAP with placebo. The primary outcome is postoperative opioid consumption measured by Patient Controlled Analgesia -pump (PCA). Secondly, subjective postoperative pain up to 24 h postoperatively will be measured by Numeric Rating Scale (NRS). Additional outcome measures are factors related to recovery and length of stay in the hospital as well as a 6 month follow-up survey regarding pain and general wellbeing after surgery. A total of 46 patients will be randomized in a proportion of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Surgery indicated because of pain caused by diagnosed or suspected peritoneal endometriosis
* ASA class 1-3
* Patient is capable of giving informed consent

Exclusion Criteria:

* Obstructive sleep apnea
* ASA class >4
* Other significant risks associated with opioid use
* Contraindications for local anesthetics or NSAIDs
* Regular opioid consumption before operation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours
  Oxicodone consumption measured via PCA-pump in Morphine equivalents

SECONDARY OUTCOMES:
Postoperative pain assessed by NRS (numeric rating scale) | Recovery room immediately postoperatively; on ward 6, 12 and 24 hours postoperatively
  NRS (numeric rating scale) with 0 (minimum) meaning no pain and 10 (maximum) meaning the worst imaginable pain
Pain at six months postoperatively; assessed by NRS (numeric rating scale), (questionnaires sent to the patients) | 6 months postop
  NRS (numeric rating scale) with 0 (minimum) meaning no pain and 10 (maximum) meaning the worst imaginable pain
Quality of life at six months postoperatively; assessed by EHP-30 (endometriosis-related health profile) (questionnaires sent to the patients) | 6 months postop
  EHP-30 (endometriosis health profile) with 0% meaning no effect on quality of life and 100% meaning maximum worsening effect on quality of life
Intra- or postoperative complications | Up to 6 months postop
  Blood loss (millilitres for each participant), Reoperation (number of participants; yes/no), Hospital stay (hours/days for each participant), Readmission (number of participants for each study group), complications according to Clavien Dindo classification (Grade I meaning any deviation from the normal postoperative course; up to grade V meaning death of patient)

CONTACTS AND LOCATIONS:
Overall Officials: Sari Koivurova, MD, PhD, Principal Investigator — Oulu University Hospital, Department of Obstetrics and Gynecology
Locations (1):
- Oulu mUniversity Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No
Anonymised data can be shared upon reasonable request to the authors.

REFERENCES:
- [Derived] Terho A, Puhto T, Laru J, Uimari O, Ohtonen P, Rautio T, Koivurova S. Laparoscopically guided transversus abdominis plane block versus local wound analgesia in laparoscopic surgery for peritoneal endometriosis: study protocol for a prospective randomized controlled double-blinded LTAP-trial. Trials. 2022 Jan 18;23(1):55. doi: 10.1186/s13063-022-06004-6. PMID 35042563